CLINICAL TRIAL: NCT04005352
Title: A 64-week, Two-arm, Randomized, Double-masked, Multicenter, Phase IIIb Study Assessing the Efficacy and Safety of Brolucizumab 6 mg Compared to Aflibercept 2 mg in a Treat-to-control Regimen in Patients With Neovascular Agerelated Macular Degeneration (TALON)
Brief Title: Study to Assess the Efficacy and Safety of Brolucizumab 6mg Compared to Aflibercept 2 mg in a Treat-to-control Regimen (TALON)
Acronym: TALON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRTH258A2303; 2019-000716-28 (EudraCT Number)
Record Dates: First submitted 2019-07-01; First posted 2019-07-02 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Age-related Macular Degeneration
Keywords: Age-related Macular Degeneration; Macular Degeneration; Wet Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases; AMD; nAMD; wet AMD; RTH258; Brolucizumab; double blind; age-related macular degeneration (ARMD); vision loss; macula damage; retina damage; dry macular degeneration; Subfoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders; Geographic Atrophy; Choroidal Neovascularization | interventions — brolucizumab; aflibercept

STUDY DESIGN:
Intervention Model Description: Double arm, multi-center
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brolucizumab 6 mg (Experimental): 3 x 4-week injections and one 8-week Intra-vitreal injection, followed by Treat-to- Control treatment from Week 16 up to Week 60/62.
  Interventions: Biological: Brolucizumab 6 mg
- Aflibercept 2 mg (Active Comparator): 3 x 4-week injections and one 8-week Intra-vitreal injection, followed by Treat-to- Control treatment from Week 16 up to Week 60/62
  Interventions: Biological: Aflibercept 2 mg

INTERVENTIONS:
Biological: Brolucizumab 6 mg — Intra-vitreal injection
  Other Names: RTH258
  Arms: Brolucizumab 6 mg
Biological: Aflibercept 2 mg — Intra-vitreal injection
  Other Names: EYLEA
  Arms: Aflibercept 2 mg

SUMMARY:
This was a 64-week randomized, double-masked, multi-center, active-controlled, two-arm study in patients with neovascular age related macular degeneration (nAMD) who have not previously received anti- vascular endothelial growth factor (VEGF) treatment.

DETAILED DESCRIPTION:
At the baseline Visit, subjects who met the eligibility criteria were randomized in a 1:1 ratio to receive either: -Brolucizumab 6 mg: 3 × 4-week injections and one 8-week injection, followed by Treat-to- Control treatment from Week 16 up to Week 60/62

-Aflibercept 2 mg: 3 × 4-week injections and one 8-week injection, followed by Treat-to-Control treatment from Week 16 up to Week 60/62.

For all subjects, the last potential study treatment was at the Week 60 visit (or at the Week 62 visit for subjects whose actual treatment interval would require a treatment at Week 62). The initiation phase starts on Day 1 and ends on Week 16. Treat to Control regimen starts on Week 16 until end of treatment (Week 60/62).

In both treatment arms, treatment intervals after the initiation phase were either 8 weeks, 12 weeks, or 16 weeks. Per the original protocol, if it was determined that a patient required more frequent injections than q8w, he/she would be moved to a q4w treatment interval. However, this option was removed per Protocol amendment 02, after which, dosing intervals shorter than q8w were not permitted.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Male or female patients ≥ 50 years of age at screening who are treatment naive
* Active choroidal neovascularization (CNV) secondary to AMD that affects the central subfield, including retinal angiomatous proliferation (RAP) with a CNV component, confirmed by presence of active leakage from CNV seen by fluorescein angiography and sequellae of CNV, e.g. pigment epithelial detachment (PED), subretinal or sub-retinal pigment epithelium (sub-RPE) hemorrhage, blocked fluorescence, macular edema (study eye)
* Presence of intraretinal fluid (IRF) or subretinal fluid (SRF) that affects the central subfield, as seen by Spectral Domain Optical Coherence Tomography (SD-OCT) (study eye)
* Best-corrected visual acuity (BCVA) score between 83 and 38 letters, inclusive, using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts at both screening and baseline visit (study eye)

Exclusion Criteria:

* Ocular conditions/disorders at screening or baseline which could, in the opinion of the investigator, prevent response to study treatment or may confound interpretation of study results, compromise visual acuity or require planned medical or surgical intervention during the first 12-month study period, structural damage of the fovea, atrophy or fibrosis at the center of the fovea (study eye)
* Any active intraocular or periocular infection or active intraocular inflammation, at screening or baseline (study eye)
* Uncontrolled glaucoma defined as intraocular pressure (IOP) > 25 mmHg on medication, or according to investigator's judgment, at screening or baseline (study eye)
* Ocular treatments: previous treatment with any anti-vascular endothelial growth factor (VEGF) drugs or investigational drugs, intraocular or periocular steroids, macular laser photocoagulation, photodynamic therapy, vitreoretinal surgery, intraocular surgery (study eye)
* Stroke or myocardial infarction during the 6-month period prior to baseline
* Systemic anti-VEGF therapy at any time.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 734 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (108):
- United States (23):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Pinellas Park, Florida
  - Novartis Investigative Site, Winter Haven, Florida
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, West Des Moines, Iowa
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Hickory, North Carolina
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Springfield, Oregon
  - Novartis Investigative Site, Germantown, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Bellaire, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
- Argentina (4):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Rosario, De Santa Fe
  - Novartis Investigative Site, Caba
- Australia (8):
  - Novartis Investigative Site, Albury, New South Wales
  - Novartis Investigative Site, Hurstville, New South Wales
  - Novartis Investigative Site, Parramatta, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Glen Waverley, Victoria
  - Novartis Investigative Site, Rowville, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Novartis Investigative Site, Vienna, Austria
- Belgium (2):
  - Novartis Investigative Site, Alken
  - Novartis Investigative Site, Leuven
- Canada (5):
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Boisbriand, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Czechia (4):
  - Novartis Investigative Site, Zlín, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Ostrava Poruba
  - Novartis Investigative Site, Prague
- France (10):
  - Novartis Investigative Site, Saint-Cyr-sur-Loire, Indre Et Loire
  - Novartis Investigative Site, Lyon, Rhone
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montauban
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rueil-Malmaison
  - Novartis Investigative Site, Strasbourg
- Germany (10):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Kempten
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Ulm
- Israel (4):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Ẕerifin
- Italy (6):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Novara
- Malaysia (3):
  - Novartis Investigative Site, Malacca, Melaka Malaysia
  - Novartis Investigative Site, Batu Caves, Selangor
  - Novartis Investigative Site, Shah Alam, Selangor
- Netherlands (2):
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Nijmegen
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Vila Franca de Xira
- South Korea (5):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Burjassot, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Zaragoza
- Sweden (2):
  - Novartis Investigative Site, Örebro
  - Novartis Investigative Site, Västerås
- Novartis Investigative Site, Binningen, Switzerland
- Taiwan (2):
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- United Kingdom (6):
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Rugby
  - Novartis Investigative Site, Sunderland
  - Novartis Investigative Site, Torquay
  - Novartis Investigative Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://clinicalstudydatarequest.com/

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1914

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 734 participants were treated.
Period: Overall Study
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Started | 366 | 368
Completed | 317 | 307
Not Completed | 49 | 61
Not completed — Adverse Event | 4 | 5
Not completed — Death | 4 | 2
Not completed — Lost to Follow-up | 6 | 2
Not completed — Physician Decision | 7 | 13
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 28 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg | Total
Number analyzed (Participants) | 366 | 368 | 734
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 37 | 69
  >=65 years | 334 | 331 | 665
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.5 (7.85) | 75.5 (8.41) | 75.5 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 204 | 420
  Male | 150 | 164 | 314
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 55 | 55 | 110
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 310 | 312 | 622
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Distribution of the Last Interval With no Disease Activity up to Week 32 - Study Eye
Description: No disease activity is defined as no change in visual acuity and no change in other signs of the disease (e.g. Intraretinal Fluid (IRF), Subretinal Fluid (SRF), hemorrhage, leakage, etc.).
  Treatment interval distribution. Number (%) of subjects at 12/8/4-weeks intervals up to Week 32 for the study eye.
  If the study treatment is discontinued before Week 16, then the treatment interval is 4 weeks; otherwise. the last interval with no disease activity is used (if there was disease activity, the last interval is shortened by 4 weeks, down to a minimum of 4 weeks).
  If the duration of the last interval falls within the following ranges of (4-week, 8-week) or (8-week, 12-week) or ≥12-week then the floor value of these ranges was used.
Time Frame: Up to Week 32
Population: Full Analysis Set (Includes participants who were randomized and treated.)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 366 | 368
Participants
  12 weeks | 141 | 73
  8 weeks | 131 | 147
  4 weeks | 94 | 148
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — with significance level of 0.025

2. Primary Outcome: Average Change From Baseline at Week 28 and Week 32 in Best-corrected Visual Acuity (BCVA) - Study Eye
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
  Least squares mean estimate - for weeks 28 and 32 combined.
Time Frame: Baseline, Week 28 and Week 32
Population: Full Analysis Set - Last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 366 | 368
Scores on a scale | 5.2 (0.51) | 5.1 (0.51)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Non-Inferiority — 4 letter margin (1-sided); p < 0.0001, ANOVA; Difference = 0.1, 95% CI 2-sided [-1.3 to 1.5], Standard Error of Mean 0.73

3. Secondary Outcome: Distribution of the Last Interval With no Disease Activity up to Week 64 - Study Eye
Description: No disease activity is defined as no change in visual acuity and no change in other signs of the disease (e.g. IRF, SRF, hemorrhage, leakage, etc.).
  Treatment interval distribution. The number of subjects at 16/12/8/4-weeks intervals as the last interval with no disease activity.
  If the study treatment is discontinued before Week 16, then the treatment interval is 4 weeks; otherwise. the last interval with no disease activity is used (if there was disease activity, the last interval is shortened by 4 weeks, down to a minimum of 4 weeks).
  If the duration of the last interval falls within the following ranges of (4-week, 8-week) or (8-week, 12-week) or (12-weeks, 16-weeks) or ≥16-week then the floor value of these ranges was used.
Time Frame: Up to Week 64
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 366 | 368
Participants
  16 Weeks | 104 | 45
  12 Weeks | 82 | 88
  8 Weeks | 95 | 81
  4 Weeks | 85 | 154
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Distribution of the Maximal Intervals With no Disease Activity up to Week 64 - Study Eye
Description: No disease activity is defined as no change in visual acuity and no change in other signs of the disease (e.g. IRF, SRF, hemorrhage, leakage, etc.).
  Maximal interval distribution. Number of subjects at 16/12/8/4-weeks intervals as the last interval with no disease activity.
  If the study treatment is discontinued before Week 16 included, then the treatment interval is 4 weeks; otherwise, the last interval with no disease activity is used (if there was disease activity, the last interval is shortened by 4 weeks, down to a minimum of 4 weeks).
  If the duration of the maximal interval falls within the following ranges of [4-weeks, 8-weeks) or [8-weeks, 12-weeks) or [12-weeks, 16-weeks] or ≥16-weeks then the floor value of these ranges is used.
Time Frame: Up to Week 64
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 366 | 368
Participants
  16 Weeks | 117 | 57
  12 Weeks | 96 | 92
  8 Weeks | 94 | 114
  4 Weeks | 59 | 105
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants With no Disease Activity - Study Eye
Description: Disease activity assessment as determined by visual acuity and assessment of other signs of the disease (e.g. IRF, SRF, hemorrhage, leakage, etc.).
Time Frame: Weeks 14 and 16
Population: Full Analysis Set. Note that the number analyzed is reduced because the Week 14 visit was conducted at the investigator's discretion, and because some patients had already stopped treatment by Week 16.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 301 | 296
Participants
  Week 14 (n=118, 137): number analyzed (Participants) | 118 | 137
  Week 14 (n=118, 137) | 87 | 88
  Week 16 (n=301,296) | 260 | 211
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 14; p = 0.0510, likelihood ratio test; Assessed at one-sided 0.025 significance level; Odds Ratio (OR) = 1.6, 95% CI 2-sided [0.9 to 2.7]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 16; p < 0.0001, likelihood ratio test; Assessed at one-sided 0.025 significance level; Odds Ratio (OR) = 2.6, 95% CI 2-sided [1.7 to 3.9]

6. Secondary Outcome: Time From Last Loading Injection to First Visit With No Disease Activity (Weeks) - 75th Percentile - Study Eye
Description: Intraretinal fluid (IRF) and subretinal fluid (SRF) were assessed by Spectral Domain Optical Coherence Tomography (SD-OCT) (study eye).
  Please note that this endpoint can be impacted by the optional disease activity assessment visits and the flexible dosing regimen, in addition to the randomized treatment. Hence, the observed treatment effect may be confounded by the study design artifacts.
Time Frame: Up to Week 64
Population: Full Analysis Set - subjects with no important protocol deviations with impact
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 366 | 368
weeks | 9.1 [8.9 to 10.6] | 12.1 [11.3 to 12.9]

7. Secondary Outcome: Time-to-first Dry Retina - Time to the First Visit With no Intraretinal Fluid (IRF) or Subretinal Fluid (SRF) - Study Eye
Description: Intraretinal fluid (IRF) and subretinal fluid (SRF) were assessed by Spectral Domain Optical Coherence Tomography (SD-OCT) (study eye).
Time Frame: Up to Week 64
Population: Full Analysis Set - subjects with no important protocol deviations with impact
Measure: Number; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 330 | 337
Participants
  0 Week | 330 | 337
  4 Week | 144 | 138
  8 Week | 70 | 86
  12 Week | 70 | 86
  16 Week | 37 | 67
  20 Week | 34 | 55
  24 Week | 30 | 47
  28 Week | 28 | 38
  32 Week | 20 | 25
  36 Week | 20 | 23
  40 Week | 18 | 22
  44 Week | 18 | 22
  48 Week | 17 | 20
  52 Week | 17 | 20
  56 Week | 17 | 20
  60 Week | 11 | 14
  64 Week | 0 | 0

8. Secondary Outcome: Average Change From Baseline at Week 60 and Week 64 in Best-corrected Visual Acuity (BCVA) - Study Eye
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
  Least squares mean estimate - for weeks 60 and 64 combined.
Time Frame: Baseline, Week 60 and Week 64
Population: Full Analysis Set - LOCF
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 366 | 368
Scores on a scale | 4.7 (0.60) | 4.9 (0.60)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; p = 0.8137, ANOVA — p-value for treatment difference; Difference = -0.2, 95% CI 2-sided [-1.9 to 1.5], Standard Error of Mean 0.84

9. Secondary Outcome: Number of Participants With Best-corrected Visual Acuity Improvements of ≥ 15 Letters in BCVA From Baseline or Reached BCVA ≥ 84 Letters up to Week 32/64 Per Treatment Arm - Study Eye
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
Time Frame: Baseline, Week 32, and Week 64
Population: Full Analysis Set - LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 366 | 368
Participants
  Week 32 | 88 | 92
  Week 64 | 89 | 91
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.4106, likelihood ratio test; adjusting for baseline BCVA categories (<55, 55-<73, ≥73 letters); Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.7 to 1.3]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.4667, likelihood ratio test; adjusting for baseline BCVA categories (<55, 55-<73, ≥73 letters); Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.7 to 1.4]

10. Secondary Outcome: Number of Participants With Best-corrected Visual Acuity ≥ 69 Letters - Study Eye
Description: as for outcome 9
Time Frame: Week 32 and Week 64
Population: Full Analysis Set - LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 366 | 368
Participants
  Week 32 | 244 | 228
  Week 64 | 240 | 219
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.2397, likelihood ratio test; assessed at the 0.025 significance level; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.8 to 1.7]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.1150, likelihood ratio test; assessed at the 0.025 significance level; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.9 to 1.8]

11. Secondary Outcome: Average Change From Baseline in Central Subfield Thickness (CSFT) - Study Eye
Description: CSFT was measured by Spectral Domain Optical Coherence Tomography
Time Frame: Baseline, Weeks 28 and 32 and at Weeks 60 and 64
Population: Full Analysis Set - LOCF
Measure: Least Squares Mean (Standard Error); unit: micrometers
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 366 | 368
micrometers
  Weeks 28 and 32 (average) | -166.9 (6.97) | -140.0 (6.96)
  Weeks 60 and 64 (average) | -182.9 (7.72) | -167.5 (8.16)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Weeks 28 and 32; p = 0.0066, ANOVA; Difference = -26.9, 95% CI 2-sided [-46.3 to -7.5], Standard Error of Mean 9.87
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Weeks 60 and 64; p = 0.1714, ANOVA; Difference = -15.4, 95% CI 2-sided [-37.6 to 6.7], Standard Error of Mean 11.26

12. Secondary Outcome: Number of Participants With Presence of Intraretinal Fluid and/or Subretinal Fluid in the Central Subfield - Study Eye
Description: Intraretinal Fluid and/or Subretinal Fluid status was measured by Spectral Domain Optical Coherence Tomography (SD-OCT).
Time Frame: At Weeks 28, 32, 60 and 64
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 286 | 289
Participants
  Week 28 (n=285,289): number analyzed (Participants) | 285 | 289
  Week 28 (n=285,289) | 175 | 198
  Week 32 (n=286, 267): number analyzed (Participants) | 286 | 267
  Week 32 (n=286, 267) | 144 | 152
  Week 60 (n=269,244): number analyzed (Participants) | 269 | 244
  Week 60 (n=269,244) | 60 | 69
  Week 64 (n=271, 241): number analyzed (Participants) | 271 | 241
  Week 64 (n=271, 241) | 72 | 83

13. Secondary Outcome: Number of Participants With Presence of Sub-Retinal Pigment Epithelium Fluid in the Central Subfield - Study Eye
Description: Sub-Retinal Pigment Epithelium fluid status was measured by Spectral Domain Optical Coherence Tomography (SD-OCT).
Time Frame: At Weeks 28, 32, 60 and 64
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 288 | 289
Participants
  Week 28 (n=288,289) | 173 | 208
  Week 32 (n=288, 266): number analyzed (Participants) | 288 | 266
  Week 32 (n=288, 266) | 156 | 175
  Week 60 (n=271,244): number analyzed (Participants) | 271 | 244
  Week 60 (n=271,244) | 27 | 31
  Week 64 (n=271, 242): number analyzed (Participants) | 271 | 242
  Week 64 (n=271, 242) | 34 | 43

14. Secondary Outcome: Change From Baseline in Visual Function Questionnnaire-25 (VFQ-25) - Composite Scores - Study Eye
Description: The National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) measures the influence of visual disability and visual symptoms on general health domains.
  The NEI VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better visual functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. Each subscale score has a range of 0 to 100 inclusive and will be calculated from the re-scaled raw data. A composite score is derived based on the average of the 11 subscales.
Time Frame: Baseline, Week 32, and Week 64
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 278 | 261
Scores on a scale
  Week 32 (n-278, 261) | 4.09 (0.20) | 3.72 (0.21)
  Week 64 (n=248, 224): number analyzed (Participants) | 248 | 224
  Week 64 (n=248, 224) | 2.8 (0.69) | 4.7 (0.73)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.193, ANCOVA; LS Mean Difference = 0.37, 95% CI 2-sided [-0.2 to 0.9]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.052, ANCOVA; LS Mean Difference = -2.0, 95% CI 2-sided [-3.9 to 0.0]

15. Secondary Outcome: Change From Baseline in Visual Function Questionnnaire-25 (VFQ-25) - Subscale Score - General Vision - Study Eye
Description: as for outcome 14
Time Frame: Baseline, Week 32, and Week 64
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 278 | 261
Scores on a scale
  Week 32 (n-278, 261) | 7.94 (0.86) | 5.79 (0.89)
  Week 64 (n=248, 224): number analyzed (Participants) | 248 | 224
  Week 64 (n=248, 224) | 7.3 (0.87) | 8.0 (0.92)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.081, ANCOVA; LS Mean Difference = 2.16, 95% CI 2-sided [-0.3 to 4.6]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.590, ANCOVA; LS Mean Difference = -0.7, 95% CI 2-sided [-3.2 to 1.8]

16. Secondary Outcome: Change From Baseline in Visual Function Questionnnaire-25 (VFQ-25) - Subscale Score - Ocular Pain - Study Eye
Description: as for outcome 14
Time Frame: Baseline, Week 32, and Week 64
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 278 | 261
Scores on a scale
  Week 32 (n-278, 261) | 3.55 (0.92) | 2.78 (0.94)
  Week 64 (n=248, 224): number analyzed (Participants) | 248 | 224
  Week 64 (n=248, 224) | 3.1 (0.89) | 5.0 (0.94)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.558, ANCOVA; LS Mean Difference = 0.77, 95% CI 2-sided [-1.8 to 3.4]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.138, ANCOVA; LS Mean Difference = -1.9, 95% CI 2-sided [-4.5 to 0.6]

17. Secondary Outcome: Change From Baseline n Visual Function Questionnnaire-25 (VFQ-25) - Subscale Score - Near Activities - Study Eye
Description: as for outcome 14
Time Frame: Baseline, Week 32, and Week 64
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 278 | 261
Scores on a scale
  Week 32 (n-278, 261) | 7.46 (1.05) | 5.86 (1.08)
  Week 64 (n=248, 224): number analyzed (Participants) | 248 | 224
  Week 64 (n=248, 224) | 4.9 (1.12) | 7.9 (1.18)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.287, ANCOVA; LS Mean Difference = 1.60, 95% CI 2-sided [-1.4 to 4.6]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.070, ANCOVA; LS Mean Difference = -3.0, 95% CI 2-sided [-6.2 to 0.2]

18. Secondary Outcome: Change From Baseline in Visual Function Questionnnaire-25 (VFQ-25) - Subscale Score - Distance Activities - Study Eye
Description: as for outcome 14
Time Frame: Baseline, Week 32, and Week 64
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 278 | 261
Scores on a scale
  Week 32 (n-278, 261) | 3.06 (0.95) | 3.78 (0.98)
  Week 64 (n=248, 224): number analyzed (Participants) | 248 | 224
  Week 64 (n=248, 224) | 2.5 (0.99) | 5.0 (1.04)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.602, ANCOVA; LS Mean Difference = -0.71, 95% CI 2-sided [-3.4 to 2.0]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.086, ANCOVA; LS Mean Difference = -2.5, 95% CI 2-sided [-5.3 to 0.4]

19. Secondary Outcome: Change From Baseline in Visual Function Questionnnaire-25 (VFQ-25) - Subscale Score - Social Functioning - Study Eye
Description: The National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) measures the influence of visual disability and visual symptoms on general health domains.
  The NEI VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better visual functioning or outcome. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. Each subscale score has a range of 0 to 100 inclusive and will be calculated from the re-scaled raw data. A composite score is derived based on the average of the 11 subscales.
Time Frame: Baseline, Week 32, and Week 64
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 278 | 261
Scores on a scale
  Week 32 (n-278, 261) | 1.99 (0.79) | 0.43 (0.82)
  Week 64 (n=247, 223): number analyzed (Participants) | 247 | 223
  Week 64 (n=247, 223) | 0.2 (0.81) | 1.7 (0.85)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.174, ANCOVA; LS Mean Difference = 1.55, 95% CI 2-sided [-0.7 to 3.8]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.210, ANCOVA; LS Mean Difference = -1.5, 95% CI 2-sided [-3.8 to 0.8]

20. Secondary Outcome: Change From Baseline in Visual Function Questionnnaire-25 (VFQ-25) - Subscale Score - Mental Health - Study Eye
Description: as for outcome 19
Time Frame: Baseline, Week 32, and Week 64
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 278 | 261
Scores on a scale
  Week 32 (n-278, 261) | 5.83 (0.99) | 6.79 (1.02)
  Week 64 (n=248, 224): number analyzed (Participants) | 248 | 224
  Week 64 (n=248, 224) | 5.0 (1.08) | 7.2 (1.14)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.499, ANCOVA; LS Mean Difference = -0.96, 95% CI 2-sided [-3.8 to 1.8]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.147, ANCOVA; LS Mean Difference = -2.3, 95% CI 2-sided [-5.4 to 0.8]

21. Secondary Outcome: Change From Baseline in Visual Function Questionnnaire-25 (VFQ-25) - Subscale Score - Role Difficulties - Study Eye
Description: as for outcome 19
Time Frame: Baseline, Week 32, and Week 64
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 278 | 261
Scores on a scale
  Week 32 (n-278, 261) | 5.17 (1.31) | 4.30 (1.35)
  Week 64 (n=248, 224): number analyzed (Participants) | 248 | 224
  Week 64 (n=248, 224) | 4.7 (1.31) | 5.9 (1.38)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.643, ANCOVA; LS Mean Difference = 0.88, 95% CI 2-sided [-2.8 to 4.6]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.507, ANCOVA; LS Mean Difference = -1.3, 95% CI 2-sided [-5.0 to 2.5]

22. Secondary Outcome: Change From Baseline in Visual Function Questionnnaire-25 (VFQ-25) - Subscale Score - Dependency - Study Eye
Description: as for outcome 19
Time Frame: Baseline, Week 32, and Week 64
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 278 | 261
Scores on a scale
  Week 32 (n-278, 261) | 2.71 (0.88) | 2.22 (0.91)
  Week 64 (n=248, 224): number analyzed (Participants) | 248 | 224
  Week 64 (n=248, 224) | -0.6 (1.09) | 2.2 (1.14)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.700, ANCOVA; LS Mean Difference = 0.49, 95% CI 2-sided [-2.0 to 3.0]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.070, ANCOVA; LS Mean Difference = -2.9, 95% CI 2-sided [-6.0 to 0.2]

23. Secondary Outcome: Change From Baseline in Visual Function Questionnnaire-25 (VFQ-25) - Subscale Score - Driving - Study Eye
Description: as for outcome 14
Time Frame: Baseline, Week 32, and Week 64
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 278 | 261
Scores on a scale
  Week 32 (n-278, 261) | 4.92 (1.56) | 4.19 (1.57)
  Week 64 (n=139, 131): number analyzed (Participants) | 139 | 131
  Week 64 (n=139, 131) | 1.3 (1.74) | 3.0 (1.79)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.741, ANCOVA; LS Mean Difference = 0.73, 95% CI 2-sided [-3.6 to 5.1]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.494, ANCOVA; LS Mean Difference = -1.7, 95% CI 2-sided [-6.6 to 3.2]

24. Secondary Outcome: Change From Baseline in Visual Function Questionnnaire-25 (VFQ-25) - Subscale Score - Color Vision - Study Eye
Description: as for outcome 14
Time Frame: Baseline, Week 32, and Week 64
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 278 | 261
Scores on a scale
  Week 32 (n-278, 261) | 1.78 (0.63) | 0.02 (0.65)
  Week 64 (n=244, 222): number analyzed (Participants) | 244 | 222
  Week 64 (n=244, 222) | 0.1 (0.80) | 1.2 (0.84)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.054, ANCOVA; LS Mean Difference = 1.76, 95% CI 2-sided [-0.0 to 3.5]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.331, ANCOVA; LS Mean Difference = -1.1, 95% CI 2-sided [-3.4 to 1.2]

25. Secondary Outcome: Change From Baseline in Visual Function Questionnnaire-25 (VFQ-25) - Subscale Score - Peripheral Vision - Study Eye
Description: as for outcome 14
Time Frame: Baseline, Week 32, and Week 64
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 278 | 261
Scores on a scale
  Week 32 (n-278, 261) | 3.24 (1.01) | 2.00 (1.04)
  Week 64 (n=243, 224): number analyzed (Participants) | 243 | 224
  Week 64 (n=243, 224) | 2.5 (1.08) | 3.0 (1.13)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 32; p = 0.394, ANCOVA; LS Mean Difference = 1.24, 95% CI 2-sided [-1.6 to 4.1]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority — Week 64; p = 0.728, ANCOVA; LS Mean Difference = -0.5, 95% CI 2-sided [-3.6 to 2.5]

26. Secondary Outcome: Number of Participants With Treatment Emergent Ocular Adverse Events (Greater Than or Equal to 1% in Any Treatment Arm) by Preferred Term for the Study Eye
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign (including abnormal laboratory findings), symptom or disease) in a subject or clinical investigation subject.
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 483 days, approx. 69 weeks, 1.3 years.
Population: Safety Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 366 | 368
Participants
  Number of subjects with at least one event | 114 | 102
  Conjunctival haemorrhage | 23 | 13
  Visual acuity reduced | 16 | 18
  Eye pain | 17 | 13
  Vitreous floaters | 12 | 6
  Intraocular pressure increased | 5 | 11
  Subretinal fluid | 5 | 11
  Vitreous detachment | 10 | 3
  Retinal haemorrhage | 4 | 7
  Cataract | 5 | 5
  Foreign body sensation in eyes | 4 | 6
  Intra-ocular injection complication | 6 | 3
  Retinal pigment epithelial tear | 5 | 4
  Macular oedema | 3 | 4
  Posterior capsule opacification | 2 | 5
  Dry eye | 2 | 4
  Hordeolum | 4 | 2
  Neovascular age-related macular degeneration | 2 | 4
  Retinal oedema | 1 | 4
  Uveitis | 4 | 1
  Vision blurred | 4 | 1
  Detachment of retinal pigment epithelium | 0 | 4
  Retinal artery occlusion | 4 | 0
  Subretinal fibrosis | 4 | 0

27. Secondary Outcome: Number of Participants With Treatment Emergent Non-ocular Adverse Events (Greater Than or Equal to 2% in Any Treatment Arm) - Summary Table
Description: as for outcome 26
Time Frame: as for outcome 26
Population: Safety Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 366 | 368
Participants | 182 | 185

ADVERSE EVENTS:
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 483 days, approx. 69 weeks, 1.3 years.
Groups:
- Brolucizumab 6mg; Aflibercept 2mg: Intra-vitreal injection
- All Patients: All Patients
Arm/Group | Brolucizumab 6mg | Aflibercept 2mg | All Patients
All-Cause Mortality (participants affected / at risk) | 4/366 | 2/368 | 6/734
Serious Adverse Events (participants affected / at risk) | 58/366 | 53/368 | 111/734
Other Adverse Events (participants affected / at risk) | 172/366 | 177/368 | 349/734
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=366) | Aflibercept 2mg (N=368) | All Patients (N=734)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 3
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 1 | 4
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1 | 3
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 1
Eye inflammation - Study Eye (Eye disorders) | 1 | 0 | 1
Glaucoma - Study Eye (Eye disorders) | 0 | 1 | 1
Iridocyclitis - Study Eye (Eye disorders) | 1 | 1 | 2
Macular hole - Study Eye (Eye disorders) | 1 | 0 | 1
Ocular discomfort - Fellow Eye (Eye disorders) | 1 | 0 | 1
Ocular discomfort - Study Eye (Eye disorders) | 1 | 0 | 1
Retinal artery occlusion - Study Eye (Eye disorders) | 1 | 0 | 1
Retinal vascular occlusion - Study Eye (Eye disorders) | 1 | 0 | 1
Retinal vein occlusion - Study Eye (Eye disorders) | 0 | 1 | 1
Uveitis - Study Eye (Eye disorders) | 3 | 0 | 3
Visual acuity reduced - Study Eye (Eye disorders) | 1 | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 0 | 2
COVID-19 pneumonia (Infections and infestations) | 5 | 1 | 6
Diverticulitis (Infections and infestations) | 0 | 2 | 2
Endophthalmitis - Study Eye (Infections and infestations) | 1 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 2
Pneumonia viral (Infections and infestations) | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1 | 3
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Intraocular pressure increased - Study Eye (Investigations) | 0 | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Basal ganglia infarction (Nervous system disorders) | 1 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Speech disorder (Nervous system disorders) | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 1
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 1 | 1 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 1
Peripheral artery aneurysm rupture (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=366) | Aflibercept 2mg (N=368) | All Patients (N=734)
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 4
Atrial fibrillation (Cardiac disorders) | 6 | 1 | 7
Vertigo (Ear and labyrinth disorders) | 4 | 4 | 8
Cataract - Study Eye (Eye disorders) | 5 | 7 | 12
Choroidal neovascularisation - Fellow Eye (Eye disorders) | 5 | 7 | 12
Conjunctival haemorrhage - Fellow Eye (Eye disorders) | 3 | 4 | 7
Conjunctival haemorrhage - Study Eye (Eye disorders) | 23 | 13 | 36
Detachment of retinal pigment epithelium - Study Eye (Eye disorders) | 0 | 4 | 4
Dry eye - Fellow Eye (Eye disorders) | 6 | 16 | 22
Dry eye - Study Eye (Eye disorders) | 8 | 18 | 26
Eye pain - Fellow Eye (Eye disorders) | 2 | 4 | 6
Eye pain - Study Eye (Eye disorders) | 17 | 13 | 30
Eye pruritus - Study Eye (Eye disorders) | 4 | 1 | 5
Foreign body sensation in eyes - Study Eye (Eye disorders) | 5 | 8 | 13
Lacrimation increased - Fellow Eye (Eye disorders) | 1 | 4 | 5
Macular oedema - Study Eye (Eye disorders) | 3 | 4 | 7
Neovascular age-related macular degeneration - Fellow Eye (Eye disorders) | 22 | 17 | 39
Neovascular age-related macular degeneration - Study Eye (Eye disorders) | 3 | 4 | 7
Posterior capsule opacification - Study Eye (Eye disorders) | 3 | 5 | 8
Retinal depigmentation - Study Eye (Eye disorders) | 1 | 4 | 5
Retinal haemorrhage - Study Eye (Eye disorders) | 4 | 7 | 11
Retinal oedema - Study Eye (Eye disorders) | 1 | 4 | 5
Retinal pigment epithelial tear - Study Eye (Eye disorders) | 5 | 4 | 9
Subretinal fibrosis - Study Eye (Eye disorders) | 4 | 0 | 4
Subretinal fluid - Study Eye (Eye disorders) | 5 | 11 | 16
Vision blurred - Study Eye (Eye disorders) | 4 | 1 | 5
Visual acuity reduced - Fellow Eye (Eye disorders) | 4 | 4 | 8
Visual acuity reduced - Study Eye (Eye disorders) | 18 | 19 | 37
Vitreous detachment - Fellow Eye (Eye disorders) | 5 | 1 | 6
Vitreous detachment - Study Eye (Eye disorders) | 11 | 3 | 14
Vitreous floaters - Study Eye (Eye disorders) | 14 | 6 | 20
Constipation (Gastrointestinal disorders) | 4 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 2 | 9
Vomiting (Gastrointestinal disorders) | 5 | 0 | 5
COVID-19 (Infections and infestations) | 9 | 16 | 25
Conjunctivitis - Fellow Eye (Infections and infestations) | 4 | 4 | 8
Conjunctivitis - Study Eye (Infections and infestations) | 5 | 5 | 10
Cystitis (Infections and infestations) | 3 | 5 | 8
Hordeolum - Study Eye (Infections and infestations) | 4 | 2 | 6
Nasopharyngitis (Infections and infestations) | 12 | 11 | 23
Urinary tract infection (Infections and infestations) | 11 | 10 | 21
Fall (Injury, poisoning and procedural complications) | 6 | 9 | 15
Intra-ocular injection complication - Study Eye (Injury, poisoning and procedural complications) | 6 | 3 | 9
Vaccination complication (Injury, poisoning and procedural complications) | 3 | 4 | 7
Gamma-glutamyltransferase increased (Investigations) | 4 | 3 | 7
Intraocular pressure increased - Study Eye (Investigations) | 5 | 10 | 15
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 1 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 6 | 10
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 8 | 16
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 2 | 8
Carpal tunnel syndrome (Nervous system disorders) | 4 | 0 | 4
Dizziness (Nervous system disorders) | 4 | 2 | 6
Headache (Nervous system disorders) | 10 | 11 | 21
Anxiety (Psychiatric disorders) | 5 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 7
Hypertension (Vascular disorders) | 18 | 17 | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT04005352/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT04005352/SAP_001.pdf